CLINICAL TRIAL: NCT04386343
Title: A Combined Phase I&II, Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate Efficacy and Safety for Prevention and Treatment of Radiation Therapy Burn of CH1701
Brief Title: CH1701 for Prevention and Treatment of Radiation Burns
Acronym: CH1701
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vietlife Healthcare Corporation (Other Government)
Collaborators: Vietnam National Cancer Hospital (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CH1701
Record Dates: First submitted 2019-08-25; First posted 2020-05-13 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase I: Three dose level - 50%, 100% and 167% of the expected dose level Phase II: Four dose level - 0% (Placebo), 50%, 100% and 167% of the expected dose level
Who Masked: Participant, Investigator
Masking Description: Participants and investigator are blinded to the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- 50% dose level arm - Phase I (Placebo Comparator): 4 healthy volunteer will use 50% dose level for Phase I in the left hand side and use placebo in the right hand side
  Interventions: Drug: Safety assessment of CH1701
- 100% dose level arm - Phase I (Placebo Comparator): 4 healthy volunteer will use 100% dose level for Phase I in the left hand side and use placebo in the right hand side
  Interventions: Drug: Safety assessment of CH1701
- 167% dose level arm - Phase I (Active Comparator): 4 healthy volunteer will use 167% dose level for Phase I in the left hand side and use placebo in the right hand side
  Interventions: Drug: Safety assessment of CH1701
- Placebo arm - Phase II (Placebo Comparator): 20 Breast cancer patients will use Placebo in the radiation affected area right after radiation
  Interventions: Drug: Placebos
- 50% dose level arm - Phase II (Placebo Comparator): 20 Breast cancer patients will use CH1701 with 50% of the expected dose level in the radiation affected area right after radiation
  Interventions: Drug: CH1701 for prevention and treatment of radiation burns.
- 100% dose level arm - Phase II (Placebo Comparator): 20 Breast cancer patients will use CH1701 with 100% of the expected dose level in the radiation affected area right after radiation
  Interventions: Drug: CH1701 for prevention and treatment of radiation burns.
- 167% dose level arm - Phase II (Placebo Comparator): 20 Breast cancer patients will use CH1701 with 167% of the expected dose level in the radiation affected area right after radiation
  Interventions: Drug: CH1701 for prevention and treatment of radiation burns.

INTERVENTIONS:
Drug: CH1701 for prevention and treatment of radiation burns. — Ch1701 is used for cancer patients who are treated with radiotherapy, then assess the safety and treatment effectiveness of the product.
  Arms: 100% dose level arm - Phase II; 167% dose level arm - Phase II; 50% dose level arm - Phase II
Drug: Safety assessment of CH1701 — Safety assessment of CH1701 after 14 days of use on volunteers
  Arms: 100% dose level arm - Phase I; 167% dose level arm - Phase I; 50% dose level arm - Phase I
Drug: Placebos — The placebo was used on patients as a control for the doses of CH1701
  Arms: Placebo arm - Phase II

SUMMARY:
A combined Phase I&II, randomized, double-blind, placebo-controlled clinical trial to evaluate efficacy and safety for prevention and treatment of radiation therapy burn of CH1701

ELIGIBILITY:
*Phase I:

Inclusion Criteria:

* Healthy volunteers, aged 18 and older at the time of enrollment
* Voluntarily participate in the study by signing a consent form to participate in the study
* Ability to adhere to treatment according to researchers' assessment

Exclusion Criteria:

* Subjects with other acute or chronic diseases need to be treated
* It is not possible to comply with the research or studied drug treatment process in the opinion of the researcher

  * Phase II:

Inclusion Criteria:

* Female patient, aged 18 to 60 years old
* Having been diagnosed with breast cancer with axillary lymph node metastasis, having radiation therapy for radiation therapy in the range of 45-50 Gy for a period of 5-6 weeks
* Treatment can be started within 3 days of signing the consent to participate in the study
* Agree to voluntarily sign the consent form to participate in the study

Exclusion Criteria:

* The available skin lesions in the breast and chest and according to the researchers' judgment will affect the assessment of inflammation caused by radiation
* The patient had radiation therapy before the breast area
* History of connective tissue disorders
* The patient is incapable of complying with the research procedures or is unable to ensure compliance with the study medication as assessed by the researcher
* Participate in other clinical trial studies within 1 month before joining this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Side effects by skin biopsy | 14 days
  Skin biopsy after 14 days of topical application, compared with healthy skin
Degree of burns according to CTCAE 4.03 atlas | 63 days
  Take photograph of skin every week comparing with atlas CTCAE 4.03 to determine the degree of burns

CONTACTS AND LOCATIONS:
Locations (1):
- Vietlife Healthcare Corporation, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided